CLINICAL TRIAL: NCT02737670
Title: Randomized Double Blind Controlled Trial on Sulodexide Efficacy in Chronic Idiopathic Subjective Tinnitus
Brief Title: Sulodexide Efficacy in Chronic Idiopathic Subjective Tinnitus
Acronym: SECIST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St Joseph University, Beirut, Lebanon (Other)
Responsible Party: Principal Investigator, Dr Joseph Maarrawi, Head of the Laboratory of Neurosciences, St Joseph University, Beirut, Lebanon
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SULO-TINNITUS
Record Dates: First submitted 2016-04-03; First posted 2016-04-14 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2017-04

CONDITIONS: Tinnitus, Subjective
MeSH Terms: conditions — Tinnitus | interventions — glucuronyl glucosamine glycan sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sulodexide (Active Comparator): Sulodexide 25 mg twice per day for 40 days
  Interventions: Drug: Sulodexide
- Placebo (Placebo Comparator): 1 tablet twice per day for 40 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sulodexide — 25 mg morning and evening for 40 days
  Arms: Sulodexide
Drug: Placebo — 1 tablet morning and evening for 40 days
  Arms: Placebo

SUMMARY:
The objective of this prospective randomized and double blind controlled study is to evaluate the efficacy and safety of Sulodexide (25 mg) in the treatment of chronic idiopathic subjective tinnitus.

DETAILED DESCRIPTION:
Patients with chronic idiopathic subjective tinnitus, since at least 1 year, re recruited from our Ear, Nose and Throat (ENT) clinic. After verification of inclusion and exclusion criteria, patients consenting to enter the study are assigned randomly to one of the following groups: 1- Sulodexide 25 mg for 40 days 2- Placebo for 40 days. Clinical evaluation of the patient is performed; tinnitus is assessed according to Tinnitus Handicap Inventory score, Mini Tinnitus Questionnaire score. Adverse effects are also noted. Patients are followed at 40 days post-treatment and outcome measures are assessed.

ELIGIBILITY:
Inclusion Criteria:

* Tinnitus for minimum of 1 year
* Absence of psychiatric or neurological diseases
* Absence of any disease that explains tinnitus
* Noise-induced hearing loss
* Cochlear and retro-cochlear damage

Exclusion Criteria:

* Conductive hearing loss
* Mixed hearing loss
* Meniere's disease
* Systemic vascular disease
* Diabetic disease
* Vestibular schwannoma
* Cerebello-pontine angle tumors
* Pulsatile tinnitus
* Pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2014-08; Primary Completion 2017-03 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Tinnitus Handicap Inventory (THI) | At day 0 and at 40 days
  Assessment of changes in THI questionnaire score between Day 40 and 0

SECONDARY OUTCOMES:
Mini Tinnitus Questionnaire (Mini-TQ) | At day 0 and at 40 days
  Assessment of changes in Mini-TQ questionnaire score between Day 40 and 0
Adverse effects | Up to 40 days
  reporting adverse effects by the patient

CONTACTS AND LOCATIONS:
Overall Officials: Elias Eter, MD, Principal Investigator — Faculty of Medicine - St Joseph University
Locations (1):
- St Jospeh University, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: Yes